CLINICAL TRIAL: NCT05108038
Title: A Randomized, Open-label, Crossover Phase 1 Clinical Trial to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety After Single/Multiple Administration of CKD-382, D860 and D027 in Healthy Subjects
Brief Title: A Study to Evaluate the PK, PD and Safety of CKD-382 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A105_02PK2115
Record Dates: First submitted 2021-10-14; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: GERD
Keywords: CKD-382; D860; D027
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- A (Experimental): Period 1: CKD-382 Period 2: D860 Period 3: D027
  Interventions: Drug: CKD-382, D860, D027
- B (Experimental): Period 1: CKD-382 Period 2: D027 Period 3: D860
  Interventions: Drug: CKD-382, D860, D027
- C (Experimental): Period 1: D860 Period 2: D027 Period 3: CKD-382
  Interventions: Drug: CKD-382, D860, D027
- D (Experimental): Period 1: D860 Period 2: CKD-382 Period 3: D027
  Interventions: Drug: CKD-382, D860, D027
- E (Experimental): Period 1: D027 Period 2: D860 Period 3: CKD-382
  Interventions: Drug: CKD-382, D860, D027
- F (Experimental): Period 1: D027 Period 2: CKD-382 Period 3: D860
  Interventions: Drug: CKD-382, D860, D027

INTERVENTIONS:
Drug: CKD-382, D860, D027 — QD, PO for 7days

SUMMARY:
to evaluate the pharmacokinetics, pharmacodynamics and safety after single/multiple administration of CKD-382, D860 and D027 in healthy subjects

DETAILED DESCRIPTION:
A randomized, open-label, crossover phase 1 clinical trial to evaluate the pharmacokinetics, pharmacodynamics and safety after single/multiple administration of CKD-382, D860 and D027 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Between 19 aged and 50 aged in healthy adult
* Body weight more than 50kg
* BMI more than 18.0 and under 27.0
* Who has negative result on Helicobacter Pylori antibody test

Exclusion Criteria:

* Have clinically significant disease that hepatobiliary system, kidney, nervous system, immune system, respiratory system, endocrine system, hemato-oncology disease, cardiovascular system or mental illness, or a history of mental disease
* Have a gastrointestinal disease history(including surgery) that can effect drug absorption
* Hypersensitivity reaction of clinically significant hypersensitivity reaction in the history of Esomeprazole, additives or benzimidazole family

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Primary Pharmacokinetic Endpoint | 0 hour(pre dose), 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours
  AUCt,ss Evaluation after multiple dose
  -AUCt,ss: Area under the plasma drug concentration-time curve within a dosing interval in steady-state
Primary Pharmacodynamic Endpoint | 24 hours after multiple dose for 7 days compared to baseline
  Percent decrease from baseline in integrated gastric acidity for 24-hour interval after 7th dose

SECONDARY OUTCOMES:
(1) Secondary Pharmacokinetic Endpoint | 0 hour(pre dose), 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours
  Cmax,ss Evaluation after multiple dose
  -Cmax,ss: Maximum concentration of drug in plasma
(1) Secondary Pharmacokinetic Endpoint | 0 hour(pre dose), 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours
  Tmax,ss Evaluation after multiple dose
  -Tmax,ss: Time to maximum plasma concentration
(1) Secondary Pharmacokinetic Endpoint | 0 hour(pre dose), 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours
  t1/2ss Evaluation after multiple dose
  -t1/ss: Terminal elimination half life in steady state
(1) Secondary Pharmacokinetic Endpoint | 0 hour(pre dose), 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours
  CLss/F Evaluation after multiple dose
  -CLss/F: Apparent Clearance in steady-state
(1) Secondary Pharmacokinetic Endpoint | 0 hour(pre dose), 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours
  Vzss/F Evaluation after multiple dose
  -Vzss/F: Apparent Volume of Distribution at steady state
(1) Secondary Pharmacokinetic Endpoint | 0 hour(pre dose), 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours
  R Evaluation after multiple dose
  -R: Accumulation ratio
(1) Secondary Pharmacokinetic Endpoint | 0 hour(pre dose), 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours
  PTF Evaluation after multiple dose
  -PTF: Peak to Trough Fluctuation
(2) Secondary Pharmacokinetic Endpoint | 0 hour(pre dose), 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours
  Cmax Evaluation after single dose
  -Cmax: Maximum concentration of drug in plasma
(2) Secondary Pharmacokinetic Endpoint | 0 hour(pre dose), 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours
  AUC0-t Evaluation after single dose
  -AUC0-t: Area under the plasma concentration-time curve from the point of administration to last time point of blood sampling
(2) Secondary Pharmacokinetic Endpoint | 0 hour(pre dose), 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours
  Tmax Evaluation after single dose
  -Tmax: Time to maximum plasma concentration
(2) Secondary Pharmacokinetic Endpoint | 0 hour(pre dose), 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours
  t1/2 Evaluation after single dose
  -t1/2: Terminal elimination half-life
(2) Secondary Pharmacokinetic Endpoint | 0 hour(pre dose), 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours
  CL/F Evaluation after single dose
  -CL/F: Apparent Clearance
(2) Secondary Pharmacokinetic Endpoint | 0 hour(pre dose), 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours
  Vz/F Evaluation after single dose
  -Vz/F: Apparent Volume of Distribution
(1) Secondary Pharmacodynamic Endpoint | 24 hours after first dose compared to baseline
  Percent decrease from baseline in integrated gastric acidity for 24-hour interval after first dose
(2) Secondary Pharmacodynamic Endpoint | 24 hours after first dose and multiple dose for 7 days
  Percent of time with gastric pH≤4 for 24-hour interval after first or 7th dose

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk Ntional University Hospital, Cheongju-si, South Korea

IPD SHARING:
Plan to Share IPD: No